CLINICAL TRIAL: NCT04146584
Title: Safety and Efficacy of SofWave Treatment to Lift Lax Tissue in the Submental and Neck Zones and to Lift the Eyebrow
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sofwave04
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Skin Laxity; Wrinkle; Brow Lifting
Keywords: Skin Laxity; Submental; Neck; Brow Lifting; Laxity; Saggy
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sofwave Treatment (Experimental): In this arm (single) patients would be treated twice with Sofwave on the face and/or submental and neck.
  Interventions: Device: Sofwave Treatments

INTERVENTIONS:
Device: Sofwave Treatments — The device used in this study will be the SofWave system manufactured by SofWave Medical ltd. The SofWave device is an ultrasonic system combined with an inherent cooling system that generates High Intensity non-focused Ultrasonic pulses (HIUS), causing a controlled thermal damage by elevating the temperature to 60-70°C in the dermis layer while sparing the epidermal layer using surface cooling. Each patient would receive 2 Sofwave treatments on the face and/or the neck.

SUMMARY:
This is a prospective, open label, multi-center, self-controlled clinical study to demonstrate the safety and efficacy of SofWave treatment to lift lax tissue in the submental and neck zones and to lift the eyebrow.

DETAILED DESCRIPTION:
This is a prospective, open label, multi-center, self-controlled clinical study to demonstrate the safety and efficacy of SofWave treatment to lift lax tissue in the submental and neck zones and to lift the eyebrow.

Up to 112 healthy candidates who are seeking treatment from participating investigators will be enrolled at up to 5 participating study sites. Patients will receive 2 treatments (4-6 weeks ± 2 weeks apart) with the SofWave system and will be followed up to 3 months post the last treatment (FU2).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between the ages 35-80.
2. Non-Smoker.
3. Fitzpatrick skin type I-VI.
4. Desire to lift lax skin in the neck and submental and/or to lift the brows.
5. Able and willing to comply with all visit, treatment and evaluation schedules and requirements.
6. Able to understand and provide written Informed Consent
7. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.
2. Presence of any active systemic or local infections.
3. Presence of active local skin disease that may alter wound healing.
4. Severe solar elastosis.
5. History of Epileptic seizures.
6. History of severe migraine tendency.
7. History of smoking in past 10 years.
8. History of chronic drug or alcohol abuse.
9. Excessive subcutaneous fat on the cheeks.
10. Significant scarring in the area to be treated.
11. Severe or cystic facial acne, acutance uses during past 6 months.
12. Presence of a metal stent or implant in the facial area.
13. Inability to understand the protocol or to give informed consent.
14. On-going use of psychiatric medication.
15. History of cosmetic treatments in the facial area to be treated, including facial skin-tightening procedure within the past year; injectable filler of any type within the past year; Botox or fillers in the lower face within the past 6 months; ablative or non-ablative resurfacing/rejuvenation laser treatment or light treatment within the past 6 months, dermabrasion or deep facial peels within the past 12 months; facelift, blepharoplasty, or brow lift (including contour threads) within the past 12 months.
16. Taking Isotretinoin or other oral retinoid within the past 6 months; taking psychiatric drugs, anti-platelet or anti-coagulant within the past 2 weeks.
17. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

    -

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Efficacy Masked Evaluators Evaluations: assessed by independent masked evaluators | 3 months post last treatment follow up visit
  Evaluate the clinical efficacy of SofWave treatment to lift lax tissue in the submental and neck zones and to lift the eyebrow, as assessed by independent masked evaluators. The two independent masked evaluators would be delivered a presentation with images randomly ordered for 'before' and 'after'. Each investigator would have to guess the correct 'after' image. Both investigators must agree on more than 50% of the cases to match success criteria. Each treated zone (Eyebrows, Neck & Submental) would be ranked individually. The primary endpoint would only be achieved along with success in outcome #5.
Safety Investigator Assessments | 3 months post last treatment follow up visit
  Evaluate the clinical safety of SofWave treatment to lift lax tissue in the submental and neck zones and to lift the eyebrow, as assessed by study physician. The investigator would examine the patient's skin before and after treatments and on follow up visits and would be requested to fill in a physician assessment, ranking Edema, erythema, ulceration/erosion, hypopigmentation and hyperpigmentation on a 5 option scale ranging from 0. - Absent to 4. Prominent. Safety would be checked every visit.

SECONDARY OUTCOMES:
Efficacy Investigator Assessments | On the second treatment visit date (pre treatment), 3 months post last treatment follow up visit
  Evaluate investigator assessment of clinical improvement in the treated zones using the Physician Global Aesthetic Improvement Scale (PGAIS). In this scale the treating physician would have to select the proper answer regarding treatment efficacy out of 5 options ranging from: 1. Very Much Improved to 5. Worse. Each treated zone (Eyebrows, Neck & Submental) would be ranked individually.
Subject Efficacy Assessments | On the second treatment visit date (pre treatment), 3 months post last treatment follow up visit
  Evaluate patient assessment of clinical improvement in the treated zones and treatment satisfaction using the patient satisfaction questionnaire. The patient would be given a patient satisfaction questionnaire with three questions regarding overall improvement (scale of 5 options ranging from 0. Worse to 4. Very much improved ), overall satisfaction (scale of 5 options ranging from 0. Very Satisfied to 4. Very Unsatisfied) and a question regarding willing to participate in future studies (options of Yes, No, Not sure). Each treated zone (Eyebrows, Neck & Submental) would be ranked individually.

OTHER OUTCOMES:
Quantitative Photo Analysis | 3 months post last follow up visit
  Photo analysis and measurements. Success criterion: point estimate of eyebrow lift > 0.5 mm Objective measurement of submental lift Success criterion: point estimate of submental lift > 20 mm. The primary endpoint would only be achieved along with success in outcome #5.

CONTACTS AND LOCATIONS:
Overall Officials: Avishai Tzur, Study Chair — Clinical Projects Manager
Locations (5):
- United States (5):
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - Laser & Skin Surgery Center of New York®, New York, New York
  - New York Laser & Skin Care, New York, New York
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Dermatology & Laser Surgery Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided